CLINICAL TRIAL: NCT07245212
Title: Testing the Efficacy of the Cannabis Clinic for Patients With Psychosis (CCP) Intervention for Cannabis Use Reduction/Cessation in Patients With First Episode Psychosis
Brief Title: Testing the Efficacy of the Cannabis Clinic for Patients With Psychosis (CCP) Intervention for Cannabis Use Reduction/Cessation in Patients With First Episode Psychosis (FEP)
Acronym: CCP RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 361577
Record Dates: First submitted 2025-11-13; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-09

CONDITIONS: Psychosis; Cannabis Use Disorder; First Episode Psychosis (FEP)
Keywords: Cannabis Use Disorder; Psychosis; First Episode Psychosis; Cannabis Cessation; Cannabis; Reduction; Cessation; Psychosocial Intervention; Psychosocial; Intervention; Cognitive Behavioural Therapy; Motivational Interviewing; Randomised Controlled Trial; Early Intervention in Psychosis; Cannabis Clinic for Psychosis; psychoeducation; peer support; flexibility; personalised
MeSH Terms: conditions — Psychotic Disorders; Marijuana Abuse | interventions — Psychosocial Intervention; Motivational Interviewing; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Waiting list single-blind RCT
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cannabis for Psychosis Intervention + Treatment as Usual (Experimental): The CCP intervention consists of two main components:
  1. one-to-one weekly sessions: offered both face to face and online to meet the patient preference. Patients can change the meeting modality at any point to suit their needs (e.g. transport difficulties, family commitments, or mental state). The CCP intervention uses a combination of evidence-based psychosocial interventions (PSIs) tailored to each patient's needs. Patients are offered on average 12 (SD 4.2) weeks sessions, for a maximum of 60 minutes
  2. an online PEER group is facilitated by a senior member of CCP staff and moderated by two PEER mentors with lived experience of psychosis and cannabis use.
  Interventions: Other: CCP Intervention
- Treatment as Usual / Waiting List (No Intervention): Participants continue Treatment as Usual from their clinical team while on a 16-week waiting list for the CCP intervention.

INTERVENTIONS:
Other: CCP Intervention — 1. one-to-one weekly sessions: offered both face to face and online to meet the patient preference. Patients can change the meeting modality at any point to suit their needs (e.g. transport difficulties, family commitments, or mental state). The CCP intervention uses a combination of evidence-based psychosocial interventions (PSIs) tailored to each patient's needs. Patients are offered on average 12 (SD 4.2) weeks sessions, for a maximum of 60 minutes.
  2. an online PEER group is facilitated by a senior member of CCP staff and moderated by two PEER mentors with lived experience of psychosis and cannabis use.
  Other Names: psychosocial intervention; motivational interviewing; cognitive behavioral therapy
  Arms: Cannabis for Psychosis Intervention + Treatment as Usual

SUMMARY:
People suffering from psychosis who use cannabis experience more relapses, long and compulsory admissions, with huge costs to the individual, families and health services. The Cannabis Clinic for Psychosis (CCP) was developed to respond to this clinical need. A published review of the CCP's intervention showed its safety and efficacy in supporting people suffering from psychosis with reducing their cannabis use. Nevertheless, for the CCP model of care to be applied widely and benefit a larger clinical population, its intervention needs to be tested in a Randomised Control Trial (RCT). The proposed CCP RCT is a waiting list randomised controlled trial that aims to evaluate the clinical efficacy of the existing CCP intervention. Participants will be adults currently under the care of South London and Maudsley (SLaM) Early Intervention Teams for first onset psychosis, who are dependent on cannabis and who express an intention to reduce or stop their use. The RCT primary outcome will measure changes in all participants' cannabis use. Participants will be randomised to either the intervention group or the waiting list control group receiving Treatment As Usual (TAU). The CCP intervention comprises 12 weekly (+/- 4 weeks) one-to-one sessions, with optional participation in a weekly online peer group. Sessions are delivered by trained clinicians and include evidence-based psychosocial techniques, including Motivational Interviewing (MI), Cognitive Behavioural Therapy (CBT), SMART goal settings and support for co-occurring tobacco use. The treatment is non-pharmacological and administered via participant-led approach that accommodates online or face-to-face sessions to meet the patient preference. Qualitative data from the recent CCP proof of concept paper indicate that the flexibility in allowing patients choice on the session's modality (online/face to face, hybrid) increased and maintained engagement.

The study is fully funded by the Maudsley Charity and due to last 30 months from the start of recruitment.

DETAILED DESCRIPTION:
Schizophrenia and other psychotic disorders are major causes of chronic ill health and early death. Daily use of high-potency cannabis significantly increases the risk of developing these disorders - up to ninefold - and also worsens outcomes and cognitive function. In the UK, it is estimated that 30-50% of patients presenting with their first episode of psychosis have been using cannabis. Approximately half of these patients continue using cannabis, and those who do are more likely to relapse, experience compulsory and longer admission hospital admissions, and experience more pronounced cognitive effects compared to those who abstain. Regardless of the clear need, there are currently few targeted interventions designed to support individuals with psychosis dependent on cannabis.

To address this urgent gap, in 2019, the first Cannabis Clinic for Psychosis (CCP) was created in the South London and Maudsley NHS Foundation Trust (SLaM) (CCP; maudsleycharity.org/case-studies/cannabis-clinic/). Cannabis use is the most modifiable risk factor for poor clinical outcomes in psychosis with strong evidence linking it to earlier illness onset, more severe symptoms and increased rates of relapse and hospitalisation. Often this population fall into two services: general adult psychiatric services or services for addiction with neither offering an intervention that addresses cannabis use directly. Despite the evidence of cannabis use having a severe impact on the outcome of people navigating psychotic disorders, there is still a lack of treatment available.

Although problematic cannabis use is becoming a significant clinical concern especially among patients with psychosis, there are currently no established treatment guidelines for this clinical population. Currently, the NICE guideline for psychosis recommends a combination of antipsychotics and general management of substance misuse, without specifically addressing the frequent co-morbidity with cannabis use disorder. This underscores a critical gap in care for individuals with psychotic disorders who are actively using cannabis while experiencing their first onset psychosis. In her Independent Review of Drugs, Professor Dame Carol Black recommended that individuals with cooccurring mental health and substance use disorders should receive integrated, concurrent treatment for both conditions. The CCP intervention offers this.

The proposed study is a waiting list randomised controlled trial (RCT) that aims to evaluate the clinical efficacy of the CCP intervention. Participants (n=80) will be adults (aged 18 and over) currently under the care of SLaM Early Intervention Teams for first onset psychosis, who are dependent on cannabis (CUDIT-R score =>9) and express an intention to reduce or stop their use. They will be randomised to either the intervention group (n=40) or the waiting list control group receiving Treatment As Usual (TAU) (N=40). The intervention comprises 12 weekly (+/- 4 weeks) one-to-one sessions, each lasting up to 60 minutes with optional participation in a weekly online peer group based on the CCP recently published proof of concept paper (POC). Sessions are delivered by trained clinicians and include evidence-based psychosocial techniques, including Motivational Interviewing (MI), Cognitive Behavioural Therapy (CBT), and personalised support for co-occurring tobacco use. The treatment is non-pharmacological and administered via participant-led approach that accommodates online or face-to-face sessions to meet the patient preference. Qualitative data from the recent CCP POC paper indicate that the flexibility in allowing patients choice on the session's modality (online/face to face, hybrid) increased and maintained engagement.

The CCP RCT primary outcome will measure, in all participants, changes in the Cannabis Use Disorders Identification Test-Revised (CUDIT-R) score between baseline (before randomisation) and at post-intervention T1 16 weeks after baseline. Other cannabis measures data will be collected at the same time points to assess pattern of use. Secondary outcomes include changes in psychosis symptoms dimensions, paranoia, depression, anxiety, cognitive and overall functioning. Previous findings from the POC analyses of the CCP intervention showed that the CUDIT-R scores, measure of Cannabis Dependence dropped from a baseline mean score 17.88 (5.15), well above the threshold for dependence (=>9) to a post intervention mean score 1.20 (2.10). 74% of participants achieved abstinence, with significant improvements across all secondary outcomes and over 90% returning to work or education. Therefore, the proposed RCT aims to formally test both the efficacy and the safety of the CCP intervention compared to a control group. Data from the CCP POC paper support an expected low risk posed to participants since the intervention is psychosocial in nature and aligned with standard care practices.

ELIGIBILITY:
Inclusion Criteria:

* First episode psychosis Community Mental Health teams receiving care under of SLaM Early Intervention for Psychosis Adult Mental Health Teams
* CUDIT≥9 (Dependent on Cannabis)
* age=18 to 65 years old ( age range of adult psychiatric services)
* Capacity to give informed consent, as assessed by clinical teams

Exclusion Criteria:

* Lack capacity to consent
* High levels of suicidal ideation, judged by clinical team

  -≥2 days/week frequency use of any other illicit drug
* Participation in any other current intervention trial
* In active crises and/or expressing suicidal ideations

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Cannabis Use Disorders Identification Test-Revised score (CUDIT-R) | Measured at a baseline assessment and 16 weeks post-randomisation.
  The CUDIT-R is an 8-item self-report tool used to screen for cannabis use and cannabis use disorder. Items assess frequency and dependence. Scores range from 0-32, with higher scores indicating greater risk.

SECONDARY OUTCOMES:
Revised Cannabis Experience Questionnaire (CEQ-mv) combined with the Enhanced cannabis timeline follow back (EC-TLFB) | Measured at a baseline assessment and 16 weeks post-randomisation.
  Self-report to assess retrospective daily cannabis use, recording weekly THC consumption in standardised units based on frequency, quantity, and potency, age of onset, potency, type, experiences and subjective effects of cannabis.
Psychotic Symptom Rating Scales Delusions Subscale (PSYRATS DEL) | Measured at a baseline assessment and 16 weeks post-randomisation.
  6-item scale designed to assess different dimensions of delusions with higher scores indicating greater symptom severity.
State Social Paranoia Scale (SSPS) | Measured at a baseline assessment and 16 weeks post-randomisation.
  10-item measure of recent paranoid thinking in a social situation with higher scores indicating greater levels of paranoia .
Patient Health Questionnaire-9 (PHQ-9) | Measured at a baseline assessment and 16 weeks post-randomisation.
  9-item measure that assesses recent levels of depression, with higher scores indicating greater levels of depression.
Generalized Anxiety Disorder-7 (GAD-7) | Measured at a baseline assessment and 16 weeks post-randomisation.
  7-item measure of assessing recent levels of anxiety, with higher scores indicating greater levels of anxiety.
Changes in the level of social activities (binary measure) | Measured at a baseline assessment and 16 weeks post-randomisation.
World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) | Measured at a baseline assessment and 16 weeks post-randomisation.
  Measures 6 domains of functioning including: cognition, mobility, self-care, getting along, life activities, participation in community
Global Assessment of Functioning (GAF) | Measured at a baseline assessment and 16 weeks post-randomisation.
  Using a scale ranging from 0 to 100, with high scores indicating no symptoms and low scores indicating impairment assessing an individual's overall psychological, social, and occupational functioning.
Days in hospital (clinical records) | Measured at a baseline assessment and 16 weeks post-randomisation.
Cannabis Withdrawal Scale (CWS) | Measured at a baseline assessment and 16 weeks post-randomisation.
  Assesses the severity of withdrawal symptoms experienced by individuals after reducing or stopping cannabis use.
Sociodemographic Schedule | Measured at a baseline assessment and 16 weeks post-randomisation.
  Includes age, gender, sex at birth, ethnicity, education, employment, marital status, living arrangements, and income source
Qualitative Questionnaire | Measured 16 weeks post-randomisation
  Assess feasibility, acceptability, and perceived impact of the CCP intervention, including barriers and facilitators to participant engagement.
Addenbrooke's Cognitive Examination (ACE) | Measured at a baseline assessment and 16 weeks post-randomisation.
  Cognitive screening tool that assesses attention, memory, language, verbal fluency, and visuospatial skills, with lower scores indicating greater cognitive impairment.
Fagerström Test for Nicotine Dependence (FTND) | Measured at a baseline assessment and 16 weeks post-randomisation.
  6-item questionnaire that measures the severity of nicotine dependence, with higher scores indicating stronger physical addiction to nicotine.

OTHER OUTCOMES:
Biological outcome | Measured at a baseline assessment and 16 weeks post-randomisation.
  Saliva cannabis drug screening test
Blood Medication levels : optional | Measured at a baseline assessment and 16 weeks post-randomisation.
  Participants will be invited to provide a sample of blood at start and end of the intervention to test if cannabis use status affects antipsychotics blood levels

CONTACTS AND LOCATIONS:
Locations (1):
- Marina House, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schoeler T, Monk A, Sami MB, Klamerus E, Foglia E, Brown R, Camuri G, Altamura AC, Murray R, Bhattacharyya S. Continued versus discontinued cannabis use in patients with psychosis: a systematic review and meta-analysis. Lancet Psychiatry. 2016 Mar;3(3):215-25. doi: 10.1016/S2215-0366(15)00363-6. Epub 2016 Jan 15. PMID 26777297
- [Background] Patel R, Wilson R, Jackson R, Ball M, Shetty H, Broadbent M, Stewart R, McGuire P, Bhattacharyya S. Association of cannabis use with hospital admission and antipsychotic treatment failure in first episode psychosis: an observational study. BMJ Open. 2016 Mar 3;6(3):e009888. doi: 10.1136/bmjopen-2015-009888. PMID 26940105
- [Background] Di Forti M, Marconi A, Carra E, Fraietta S, Trotta A, Bonomo M, Bianconi F, Gardner-Sood P, O'Connor J, Russo M, Stilo SA, Marques TR, Mondelli V, Dazzan P, Pariante C, David AS, Gaughran F, Atakan Z, Iyegbe C, Powell J, Morgan C, Lynskey M, Murray RM. Proportion of patients in south London with first-episode psychosis attributable to use of high potency cannabis: a case-control study. Lancet Psychiatry. 2015 Mar;2(3):233-8. doi: 10.1016/S2215-0366(14)00117-5. Epub 2015 Feb 25. PMID 26359901
- [Background] Lin J, Puigserver P, Donovan J, Tarr P, Spiegelman BM. Peroxisome proliferator-activated receptor gamma coactivator 1beta (PGC-1beta ), a novel PGC-1-related transcription coactivator associated with host cell factor. J Biol Chem. 2002 Jan 18;277(3):1645-8. doi: 10.1074/jbc.C100631200. Epub 2001 Nov 30. PMID 11733490